CLINICAL TRIAL: NCT04158661
Title: Influence of Minimally Invasive Thymectomy on the Subsequent Clinical Course of Myasthenia Gravis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other); Department of Surgery, Charite, Berlin (Unknown); Sana Klinikum Lichtenberg, Berlin (Unknown)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: Mya-Thymektomie
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Robotic-assisted minimally-invasive thymectomy; Mean daily prednisone dose
MeSH Terms: conditions — Myasthenia Gravis | interventions — Thymectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tmin-group: * confirmed seropositive ocular or generalized MG [detection of antibodies (Abs) targeting the AChR, muscle-specific tyrosine kinase (MuSK) or Titin] or seronegative ocular or generalized MG
  * age ≥ 18 years
  * thymectomy ≥ three years
  Interventions: Procedure: thymectomy (robotic-assisted thoracoscopic, minimally-invasive thymectomy)
- T0-group: * confirmed seropositive ocular or generalized MG [detection of antibodies (Abs) targeting the AChR, muscle-specific tyrosine kinase (MuSK) or Titin] or seronegative ocular or generalized MG
  * a very long disease history OR
  * age ≥ 18 years
  * rejecting a thymectomy or have contraindications for thymectomy
  Interventions: Procedure: no thymectomy (control)
- MGTX-group ("historical control group"): from MGTX-trial ("Randomized Trial of Thymectomy in Myasthenia Gravis")
  Interventions: Procedure: thymectomy by means of median sternotomy (transsternal)

INTERVENTIONS:
Procedure: thymectomy (robotic-assisted thoracoscopic, minimally-invasive thymectomy) — preferring one unilateral access and placing three trocars between 3rd and 5th intercostal space in a triangular configuration, with a goal of an en bloc resection of all mediastinal tissue that could anatomically contain gross or microscopic thymus (or both).
  Groups: Tmin-group
Procedure: thymectomy by means of median sternotomy (transsternal) — with a goal of an en bloc resection of all mediastinal tissue that could anatomically contain gross or microscopic thymus (or both).
  Groups: MGTX-group ("historical control group")
Procedure: no thymectomy (control) — routine medical care
  Groups: T0-group

SUMMARY:
The aim of this study is to investigate whether minimally invasive thymectomy achieves comparable efficacy and safety results compared to open thymectomy in patients with myasthenia gravis. The planned investigation is a multicenter observational study based on retrospective (present patient data) and prospective data (questionable outcome data).

Primary hypothesis: Minimally invasive thymectomy is not inferior to open thymectomy in terms of efficacy and safety (non-inferiority study).

DETAILED DESCRIPTION:
Based on large cohort studies of the last decades, the thymectomy has become a central component of the immunomodulating therapy in MG patients without thymoma detection. Because randomized studies were missing, remained a residual uncertainty on the importance of Thymectomy. In the study "Randomized Trial of Thymectomy in Myasthenia Gravis" (MGTX-study) published 2016 the effectiveness of thymectomy by patients without thymoma detection has been indisputable confirmed. A significant improvement of the patient's complaints and the reduction of the immunosuppressive drugs were particularly evident by early onset MG (EOMG) two to three years after performing a complete resection of the thymic tissue.

While the MGTX study (with an open operative procedure) was being done, the minimally-invasive thymectomy has gained more and more acceptance. From a surgical point of view, the minimally invasive thoracoscopic procedure represents a gentler alternative. According to the momentaneous clinical-scientific point of view, further studies are necessary to compare both procedures. Furthermore, the MGTX study included only patients with generalized MG and positive anti-Acetylcholine Receptor (AChR)-antibodies, who were younger than 65 years, so that the relevance of thymectomy in other important subgroups, such as late onset MG (LOMG), the ocular MG (OMG), as well as the patients without detected antibodies (seronegative MG patients), who represent about 10 % of whole population of MG patients, is still not clear.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Myasthenia Gravis
* Age ≥18 years

Exclusion Criteria:

* a proper communication with the patient is not possible
* an informed consent could not be signed
* a patient reject a participation or requires breaking up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of myasthenia gravis by:
  * typical clinical features AND
  * antibody diagnostic AND
  * positive edrophonium test OR
  * abnormal repetitive nerve stimulation OR
  * abnormal single-fiber electromyography.
  Myasthenia Gravis Foundation of America clinical classification (MGFA classification) of I to V was accepted (class I indicates weakness only in ocular muscles, class II mild generalized disease, class III moderate generalized disease, class IV severe generalized disease and class V a crisis requiring Intubation)
  Participants could be taking appropriate anticholinesterase therapy with or without oral glucocorticoids
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean daily prednisone dose | three years after thymectomy

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, Prof. Dr. med., Principal Investigator — Charité University, Berlin, Germany
Locations (3):
- Germany (3):
  - Sana Klinikum Lichtenberg, Berlin
  - Department of Surgery Charité University, Mitte
  - NeuroCure Clinical Research Center (NCRC), Charité University, Berlin, Mitte

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolfe GI, Kaminski HJ, Aban IB, Minisman G, Kuo HC, Marx A, Strobel P, Mazia C, Oger J, Cea JG, Heckmann JM, Evoli A, Nix W, Ciafaloni E, Antonini G, Witoonpanich R, King JO, Beydoun SR, Chalk CH, Barboi AC, Amato AA, Shaibani AI, Katirji B, Lecky BR, Buckley C, Vincent A, Dias-Tosta E, Yoshikawa H, Waddington-Cruz M, Pulley MT, Rivner MH, Kostera-Pruszczyk A, Pascuzzi RM, Jackson CE, Garcia Ramos GS, Verschuuren JJ, Massey JM, Kissel JT, Werneck LC, Benatar M, Barohn RJ, Tandan R, Mozaffar T, Conwit R, Odenkirchen J, Sonett JR, Jaretzki A 3rd, Newsom-Davis J, Cutter GR; MGTX Study Group. Randomized Trial of Thymectomy in Myasthenia Gravis. N Engl J Med. 2016 Aug 11;375(6):511-22. doi: 10.1056/NEJMoa1602489. PMID 27509100